CLINICAL TRIAL: NCT05300035
Title: A Randomised Phase II Placebo-controlled Trial of Antiretroviral Therapy (ART) Plus Dual Long-acting HIV-specific Broadly Neutralising Antibodies (bNAbs) vs ART Plus Placebo During Primary HIV-1 Infection to Study the Impact on Post-treatment HIV Control.
Brief Title: Phase II Trial of ART + Dual bNAbs vs. ART + Placebo During Primary HIV-1 Infection-impact on Post-ART Control
Acronym: RHIVIERA-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Rockefeller University (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANRS 176 RHIVIERA-02
Record Dates: First submitted 2022-01-03; First posted 2022-03-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: HIV/AIDS and Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — Broadly Neutralizing Antibodies; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bNAbs (Active Comparator): ART plus dual long-acting (LS) broadly neutralising antibodies (bNAbs) infusion at HIV-1 primary HIV-1 infection, during 52 weeks minimum, followed by and Antiretroviral Treatment Interruption (ATI).
  Interventions: Drug: Recombinant human monoclonal antibody (bNAbs)
- Placebo (Placebo Comparator): ART plus placebo (saline solution) at HIV-1 primary HIV-1 infection, during 52 weeks minimum, followed by and Antiretroviral Treatment Interruption (ATI).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant human monoclonal antibody (bNAbs) — 1. Initiation of combination ART (1 integrase inhibitor + 2 nucleoside analogue reverse transcriptase inhibitors) with additional dual intravenous infusions of bNAbs (3BNC117LS & 10-1074LS) between Day 7 and Day 10.
  2. Analytical treatment interruption (ATI), 52 weeks later, if good immunologic and virologic conditions.
  3. During ATI, plasma HIV-1 RNA and CD4 monitoring, for a maximum of 48 weeks.
  4. ART resumption, if participant encounters at least one ART resumption criteria.
  Other Names: 10-1074-LS and 3BNC117-LS
  Arms: bNAbs
Drug: Placebo — 1. Initiation of combination ART (1 integrase inhibitor + 2 nucleoside analogue reverse transcriptase inhibitors) with additional dual intravenous infusions of placebo (saline solution) between Day 7 and Day 10.
  2. Analytical treatment interruption (ATI), 52 weeks later, if good immunologic and virologic conditions.
  3. During ATI, plasma HIV-1 RNA and CD4 monitoring, for a maximum of 48 weeks.
  4. ART resumption, if participant encounters at least one ART resumption criteria.
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
RHIVIERA-02 trial is a placebo-controlled double-blinded two arm prospective phase II trial. This study will test the use of broadly neutralising antibodies (bNAbs) in participants, at primary HIV infection (PHI) and ART initiation.

DETAILED DESCRIPTION:
The study proposes to test an intervention consisting of dual long-acting HIV-specific broadly neutralizing antibodies (3BNC117-LS & 10-1074-LS ) + ART, at primary HIV-1 infection, and to compare it to ART only regarding HIV-1 replication.

The study aims to enrol 69 participants in French (Ile-de-France) clinical centres. Participants will have been diagnosed with primary HIV-1 infection, will start ART during early phase of Primary HIV infection, and will interrupt ART 52 weeks later.

Study duration will vary by participant, depending on the time of ART interruption and the time to viral rebound.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary HIV-1 infection diagnostic
* Aged ≥18 to ≤70 years old at screening
* Willing to use use an effective method of contraception from the inclusion until the end of the follow-up in the trial
* Negative plasmatic beta human chorionic gonadotropin (β-HCG) pregnancy test, when applicable
* Agree not to seek pregnancy including through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit, when applicable
* Informed and written signed consent
* Participant with regular health insurance
* Willing to accept the trial constraints (travel for IMP administration and ART interruption)
* Willing to be vaccinated against COVID-19 according to recommandations

Exclusion Criteria:

* Participation in any other clinical trial requiring additional blood sampling Participation in an observational study without additional blood sampling is permitted
* Participants in whom condom use or PrEP use by the partner will be difficult or impossible
* Pregnant or breastfeeding patient
* Participants under guardianship or curatorship
* Any condition or infection, including HCV, HBV, SARS-CoV-2 or known M. tuberculosis active infection History of ischemic heart disease (myocardial infarction, stable or unstable angina, stroke)
* Current or past history of cancer, excluding squamous cell skin cancers
* History or acute known inflammatory ophthalmic affection (uveitis, choroiditis, optic neuropathy)
* Any medical condition that contraindicates ART interruption
* Concomitant or previous conditions that preclude injection of monoclonal antibodies
* History of systemic corticosteroids, immunosuppressive and anti-cancer medications within the last 6 months
* History of severe reaction to a vaccine or drug infusion or history of severe allergic reactions
* Individuals with any contraindication (including hypersensitivity reaction) to 3BNC117-LS and 10-1074-LS infusion
* Prothrombin < 50%
* Creatinine clearance < 60mL/mn (Cockroft)
* ASAT or ALAT or bilirubine (total et conjugated) ≥ 10 times the upper limit of normal
* Patient with an isolated HIV-2 viral strain
* Planned absence that could affect participation in the trial (travel abroad, relocation, impending transfer...)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2028-12-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with plasma HIV-1 RNA below 400 cp/mL 24 weeks following ATI (W24 ATI), in the confirmed absence of ART. | at Week 24 of antiretroviral treatment interruption period (ATI)
  These participants will be considered as post-treatment controllers.

SECONDARY OUTCOMES:
Tolerance of bNAbs infusion : Number of clinical and biological adverse event (AE) | from date of inclusion to the last follow-up visit date, up to 148 weeks
  Number of clinical and biological AE during follow-up. Abnormal laboratory values will be identified as those outside values defined by the DAIDS scale
Tolerance of bNAbs infusion : Nature and Grade of clinical and biological AE | from date of inclusion to the last follow-up visit date, up to 148 weeks
  Grade of clinical and biological adverse during follow-up. The intensity of all AE (serious and non-serious) will be graded using the DAIDS AE Grading Table Corrected Version 2.1-July 2017
Tolerance of bNAbs infusion : Time of clinical and biological adverse event (AE) | from date of inclusion to the last follow-up visit date, up to 148 weeks
Proportion of participants resuming ART within the first 24 weeks of ART interruption, according to the reason for resuming. | at Week 24 of antiretroviral treatment interruption period (ATI)
Time to potential ART resumption for non-controllers. | from Day 0 of antiretroviral treatment interruption period (ATI) to Day 0 of ART resumption date, assessed up to 48 weeks following ATI
Clinical and immulogical criteria during follow-up: Proportion of participants with clinical symptoms. | during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
Clinical and immulogical criteria during follow-up: Evolution of CD4, CD8 (levels and %) and CD4/CD8 ratio. | during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
Clinical and immulogical criteria during follow-up: Evolution of inflammation markers levels. | biological parameters levels during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
  physiological parameters levels will be studied: IP10, TGFβ, IL-7, IL-10, IL-12, IL-15, IL-18, Citrulline, sCD14, sCD163, TNF-α
Immulogical criteria : Changes in the magnitude and quality of HIV-specific T cell responses and humoral responses. | physiological parameters levels during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
  physiological parameters levels will be studied: frequency and functionality of T cells responding to HIV peptides measured by intracellular cytokine staining, surface expression of activation and differentiation markers, HIV suppressive capacity upon co-culture with autologous infected cells
Virological criteria during follow-up: Plasma HIV-1 RNA and HIV-1 DNA level and cell-associated HIV RNA transcripts changes. | during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
Virological criteria : Proportion of participant with plasma HIV-1 RNA < 50 cp/mL at 12- and 24-weeks following ART interruption. | at Week 12 and Week 24 of antiretroviral treatment interruption period (ATI)
Virological criteria : Cumulative plasma viremia during ART interruption. | from Day 0 of antiretroviral treatment interruption period (ATI) to Day 0 of ART resumption, assessed up to 48 weeks following ATI
Virological criteria : in case of ART resumption, time from date of ART interruption begining to date of first HIV-1 RNA ≥ 50 copies/mL | from Day 0 of antiretroviral treatment interruption period (ATI) to Day 0 of ART resumption, assessed up to 48 weeks following ATI
Virological criteria : in case of ART resumption, proportion of participant with plasma HIV-1 RNA < 50 copies/mL within 24 weeks of ATI. | from Day 0 of antiretroviral treatment interruption period (ATI) to Day 0 of ART resumption, assessed up to 48 weeks following ATI
Virological criteria : Evolution of total HIV-1 DNA and cell-associated HIV-1 RNA by US q-PCR and predictive value on post- ART interruption evolution. | during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
Virological criteria : Evolution of detection proportion and level of cell-associated HIV-1 RNA. | during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
Virological criteria : Qualitative and quantitative changes in the persistent viral reservoir. | physiological parameters levels during all ART period (from Day 0 to Week 52 ARV), during all ATI period (from Day 0 ATI to Day 0 ART Resumption) and during ART resumption period (from Day 0 to Week 24 ART Resumption)
  physiological parameters levels will be studied: total cell associated HIV-DNA, integrated HIV-DNA, proportion of replication competent vs defective proviruses
Dosages of bNAbs performed during follow-up. | during ART follow-up (Week 1,Week 12, Week 24, Week 36), and antiretroviral treatment interruption period (Day 0, Week 12, Week 24)
Criteria related to the risk of HIV-1 transmission : Proportion of participants reporting to use condoms during sexual intercourses | from date of inclusion to the last follow-up visit date, up to 148 weeks
Criteria related to the risk of HIV-1 transmission : Proportion of participants reporting to have proposed PrEP at their partners. | from date of inclusion to the last follow-up visit date, up to 148 weeks
Social sciences criteria : Proportion of patients satisfied with their participation and the associated factors | from date of inclusion to the last follow-up visit date, up to 148 weeks
Social sciences criteria : Impact of the participation in the trial on participant quality of life and quality of sexual life | from date of inclusion to the last follow-up visit date, up to 148 weeks
  Through statistical analyses of some self-administered questionnaires items (in particular the SF12.v2 scale for quality of life) and thematic analyses of semi-directive individual interviews we will highlight the impact of the participation in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Goujard, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (17):
- France (17):
  - Hôpial Avicenne - SMIT, Bobigny
  - Hôpital Antoine Béclère, Clamart
  - Hôpital Beaujon - Service de médecine interne, Clichy
  - CHI Créteil - HdJ, Créteil
  - Hôpital Raymond Poincaré - SMIT, Garches
  - Hôpital Bicêtre - HdJ - Médecine interne, Le Kremlin-Bicêtre
  - Hôpital Hôtel - Dieu, Paris
  - Hôpital Hôtel Dieu - Service d'immunologie clinique, Paris
  - Hôpital Pitié-Salpêtrière - SMIT, Paris
  - Hôpital Lariboisière - Service de médecine interne A, Paris
  - Hôpital Saint- Louis - SMIT, Paris
  - Hôpital Saint-Antoine - SMIT, Paris
  - Hôpital Necker - SMIT, Paris
  - Hôpital Bichat - Claude Bernard - SMIT, Paris
  - Hôpital Tenon - SMIT, Paris
  - Centre médico chirurgical Foch - Suresnes, Suresnes
  - CHI Villeneuve-Saint-Georges - SMIT, Villeneuve-Saint-Georges